CLINICAL TRIAL: NCT03350737
Title: Coronary ARteriogenesis With Combined Heparin and EXercise Therapy in Chronic Refractory Angina
Brief Title: Coronary Arteriogenetic Heparinized Exercise
Acronym: CARHEXA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Centre of Serbia (Other)
Collaborators: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Responsible Party: Principal Investigator, Branko Beleslin, Clinical research, Clinical Centre of Serbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 128/8
Record Dates: First submitted 2017-11-08; First posted 2017-11-22 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Refractory Angina; Chronic Stable Angina
Keywords: No-option patients
MeSH Terms: conditions — Angina Pectoris; Angina, Stable | interventions — Heparin; Protons

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open-label study design. These "no-option" patients will be allocated (16 for each group) to 2 treatments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heparin-primed physical rehabilitation (Experimental): 2 exercise sessions per day for 5 days a week for 2 weeks with 100 IU/kg of Heparin i.v. (up to a maximum of 5000 IU) 10 minutes prior to exercise
  Interventions: Other: Physical rehabilitation; Drug: Heparin
- Placebo-primed physical rehabilitation (Placebo Comparator): 2 exercise sessions per day for 5 days a week for 2 weeks with placebo (2 ml of Sodium Chloride 0.9% i.v.) 10 minutes prior to exercise
  Interventions: Other: Physical rehabilitation; Other: Placebo

INTERVENTIONS:
Other: Physical rehabilitation — Standard treadmill exercise session
  Other Names: E
Drug: Heparin — Heparin i.v.
  Other Names: H
  Arms: Heparin-primed physical rehabilitation
Other: Placebo — Sodium Chloride 0.9% i.v.
  Other Names: P
  Arms: Placebo-primed physical rehabilitation

SUMMARY:
This study evaluates the addition of heparin to a 2-week cycle of physical rehabilitation in the treatment of refractory angina. Half of the patients will undergo heparin-primed physical rehabilitation, while the other half will undergo only physical rehabilitation.

DETAILED DESCRIPTION:
Our approach is based on the combination of pharmacological stimuli (with heparin) on top of a 2-week cycle of physical rehabilitation. The rationale for this chemical-physical cocktail stems from the fact that increase in shear stress (achieved with exercise), or heparin (when used alone) have no significant effect on coronary arteriogenesis. Nevertheless, when the two stimuli are coupled coronary arteriogenesis is consistently present, and clinically significant.

The basic principle of heparin treatment is to potentiates angiogenic growth factors, which are over expressed by increased shear stress at the site of pre-existing collateral vessels as a result of exercise or pacing. Although the precise mechanisms by which heparin potentiates arteriogenesis remain to be completely elucidated, heparin administration combined with exercise has great potential in treating patients with effort angina who are not indicated for conventional revascularization therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented coronary artery disease not amenable of future treatment and belonging to "no-option" category with symptoms consistent with angina pectoris

Exclusion Criteria:

* Patients with unstable angina, recent myocardial infarction, uncontrolled hypertension, hemodynamically valvular heart disease, bronchial asthma, and neurologic and/or orthopedic illnesses that limit exercise capacity .
* Patients receiving vitamin K antagonist.
* Patients actively involved in programmes of cardiac rehabilitation or exercise training.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Canadian Cardiovascular Society (CCS) angina severity class at 2 weeks | 2 weeks
  CCS class ranging from 1 (mild) to 4 (severe) before and after the 2-week physical rehabilitation.

SECONDARY OUTCOMES:
Change from Baseline peak stress wall motion score index (WMSI) at 2 weeks | 2 weeks
  Peak WMSI at stress echocardiography before and after 2-week physical rehabilitation at . Wall motion score index is assessed by using 17- segment model of left ventricle (1=normal, 4=dyskinetic).
Change from baseline peak stress global longitudinal strain (GLS) at 2 weeks | 2 weeks
  Peak stress GLS assessed by echocardiography before and after the 2-week physical rehabilitation.

OTHER OUTCOMES:
Change from Baseline Coronary Collateral Circulation (CCC) at 2 weeks | 2 weeks
  CCC score assessed by multi dimensional computed tomography (CT) before and after 2-week physical rehabilitation. Distal filling of the epicardial segment is semiquantitatively classified by using a four-point scale according to patterns at coronary CT angiography (CTA) (0 = absence of distal filling; 1 = partial distal filling, with a length less than one-third of the segment; 2 = partial distal filling, with a length between one-third and two-thirds of the segment; 3 = complete or partial distal filling, with a length longer than two-thirds of the segment). A coronary CTA scores correspond fully to Rentrop classification (coronary CTA score of 0 or 1 to Rentrop 0 or 1, coronary CTA score of 2 or 3 to Rentrop 2 or 3). Coronary CTA score of 3 is indicative of well-developed collaterals, contrary to scores of 0-2 (poorly developed). Also we look for change in growth of baseline bridging antegrade collaterals at 2 weeks (0= not present, 1= present)
Change from Baseline Stable Angina questionnaire (SAQ) at 4 weeks | 2 weeks to one month
  19-item Seattle SAQ that assesses angina frequency, angina stability, physical limitations, treatment satisfaction, and disease perception/QoL

CONTACTS AND LOCATIONS:
Overall Officials: Branko Beleslin, MD, PhD, Principal Investigator — Clinical Centre of Serbia; Ana Djordjevic-Dikic, MD, PhD, Study Director — Clinical Centre of Serbia; Eugenio Picano, MD, PhD, Study Chair — Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy
Locations (1):
- Clinical Centre of Serbia, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP
Time Frame: After the study completion.
Access Criteria: For collaborators, data analyses upon request.

REFERENCES:
- [Background] Barron HV, Sciammarella MG, Lenihan K, Michaels AD, Botvinick EH. Effects of the repeated administration of adenosine and heparin on myocardial perfusion in patients with chronic stable angina pectoris. Am J Cardiol. 2000 Jan 1;85(1):1-7. doi: 10.1016/s0002-9149(99)00596-2. PMID 11078227
- [Background] Bolognese L, Carrabba N, Parodi G, Santoro GM, Buonamici P, Cerisano G, Antoniucci D. Impact of microvascular dysfunction on left ventricular remodeling and long-term clinical outcome after primary coronary angioplasty for acute myocardial infarction. Circulation. 2004 Mar 9;109(9):1121-6. doi: 10.1161/01.CIR.0000118496.44135.A7. Epub 2004 Feb 16. PMID 14967718
- [Background] Bombardini T, Picano E. The coronary angiogenetic effect of heparin: experimental basis and clinical evidence. Angiology. 1997 Nov;48(11):969-76. doi: 10.1177/000331979704801106. PMID 9373049
- [Background] Buschmann I, Schaper W. Arteriogenesis Versus Angiogenesis: Two Mechanisms of Vessel Growth. News Physiol Sci. 1999 Jun;14:121-125. doi: 10.1152/physiologyonline.1999.14.3.121. PMID 11390835
- [Background] Fujita M, Sasayama S, Asanoi H, Nakajima H, Sakai O, Ohno A. Improvement of treadmill capacity and collateral circulation as a result of exercise with heparin pretreatment in patients with effort angina. Circulation. 1988 May;77(5):1022-9. doi: 10.1161/01.cir.77.5.1022. PMID 2834115
- [Background] Gibbons RJ, Abrams J, Chatterjee K, Daley J, Deedwania PC, Douglas JS, Ferguson TB Jr, Fihn SD, Fraker TD Jr, Gardin JM, O'Rourke RA, Pasternak RC, Williams SV, Gibbons RJ, Alpert JS, Antman EM, Hiratzka LF, Fuster V, Faxon DP, Gregoratos G, Jacobs AK, Smith SC Jr; American College of Cardiology; American Heart Association Task Force on Practice Guidelines. Committee on the Management of Patients With Chronic Stable Angina. ACC/AHA 2002 guideline update for the management of patients with chronic stable angina--summary article: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee on the Management of Patients With Chronic Stable Angina). Circulation. 2003 Jan 7;107(1):149-58. doi: 10.1161/01.cir.0000047041.66447.29. No abstract available. PMID 12515758
- [Background] Mannheimer C, Camici P, Chester MR, Collins A, DeJongste M, Eliasson T, Follath F, Hellemans I, Herlitz J, Luscher T, Pasic M, Thelle D. The problem of chronic refractory angina; report from the ESC Joint Study Group on the Treatment of Refractory Angina. Eur Heart J. 2002 Mar;23(5):355-70. doi: 10.1053/euhj.2001.2706. No abstract available. PMID 11846493
- [Background] Meier P, Gloekler S, de Marchi SF, Indermuehle A, Rutz T, Traupe T, Steck H, Vogel R, Seiler C. Myocardial salvage through coronary collateral growth by granulocyte colony-stimulating factor in chronic coronary artery disease: a controlled randomized trial. Circulation. 2009 Oct 6;120(14):1355-63. doi: 10.1161/CIRCULATIONAHA.109.866269. Epub 2009 Sep 21. PMID 19770393
- [Background] Picano E, Alaimo A, Chubuchny V, Plonska E, Baldo V, Baldini U, Pauletti M, Perticucci R, Fonseca L, Villarraga HR, Emanuelli C, Miracapillo G, Hoffmann E, De Nes M. Noninvasive pacemaker stress echocardiography for diagnosis of coronary artery disease: a multicenter study. J Am Coll Cardiol. 2002 Oct 2;40(7):1305-10. doi: 10.1016/s0735-1097(02)02157-5. PMID 12383579
- [Background] Picano E, Michelassi C. Chronic oral dipyridamole as a 'novel' antianginal drug: the collateral hypothesis. Cardiovasc Res. 1997 Mar;33(3):666-70. doi: 10.1016/s0008-6363(96)00262-3. PMID 9093537
- [Background] Picano E; PISA (Persantin In Stable Angina) study group. Dipyridamole in chronic stable angina pectoris; a randomized, double blind, placebo-controlled, parallel group study. Eur Heart J. 2001 Oct;22(19):1785-93. doi: 10.1053/euhj.2001.2623. PMID 11549300
- [Background] Rentrop KP, Cohen M, Blanke H, Phillips RA. Changes in collateral channel filling immediately after controlled coronary artery occlusion by an angioplasty balloon in human subjects. J Am Coll Cardiol. 1985 Mar;5(3):587-92. doi: 10.1016/s0735-1097(85)80380-6. PMID 3156171
- [Background] Schirmer SH, van Nooijen FC, Piek JJ, van Royen N. Stimulation of collateral artery growth: travelling further down the road to clinical application. Heart. 2009 Mar;95(3):191-7. doi: 10.1136/hrt.2007.136119. PMID 19144878
- [Background] Sicari R, Nihoyannopoulos P, Evangelista A, Kasprzak J, Lancellotti P, Poldermans D, Voigt JU, Zamorano JL; European Association of Echocardiography. Stress Echocardiography Expert Consensus Statement--Executive Summary: European Association of Echocardiography (EAE) (a registered branch of the ESC). Eur Heart J. 2009 Feb;30(3):278-89. doi: 10.1093/eurheartj/ehn492. Epub 2008 Nov 11. No abstract available. PMID 19001473
- [Background] Tateno S, Terai M, Niwa K, Jibiki T, Hamada H, Yasukawa K, Honda T, Oana S, Kohno Y. Alleviation of myocardial ischemia after Kawasaki disease by heparin and exercise therapy. Circulation. 2001 May 29;103(21):2591-7. doi: 10.1161/01.cir.103.21.2591. PMID 11382729
- [Background] Traupe T, Gloekler S, de Marchi SF, Werner GS, Seiler C. Assessment of the human coronary collateral circulation. Circulation. 2010 Sep 21;122(12):1210-20. doi: 10.1161/CIRCULATIONAHA.109.930651. No abstract available. PMID 20855668
- [Background] Williams B, Menon M, Satran D, Hayward D, Hodges JS, Burke MN, Johnson RK, Poulose AK, Traverse JH, Henry TD. Patients with coronary artery disease not amenable to traditional revascularization: prevalence and 3-year mortality. Catheter Cardiovasc Interv. 2010 May 1;75(6):886-91. doi: 10.1002/ccd.22431. PMID 20432394
- [Background] Wykrzykowska JJ, Henry TD, Lesser JR, Schwartz RS. Imaging myocardial angiogenesis. Nat Rev Cardiol. 2009 Oct;6(10):648-58. doi: 10.1038/nrcardio.2009.157. Epub 2009 Sep 8. PMID 19736553

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-12-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT03350737/Prot_SAP_000.pdf